CLINICAL TRIAL: NCT06732193
Title: Clinical Trial Comparing a Face-to-face Perioperative Respiratory Physiotherapy Program Versus the Use of Fissios App© as a Complement to a Respiratory Physiotherapy Program in Patients Diagnosed With NSCLC Undergoing Surgery.
Brief Title: Fissios© and Postoperative Complications (FPoC Trial)
Acronym: FPoC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Carlos Alfredo Fraile Olivero, MD, PhD. (Other)
Collaborators: Spanish Society of Pneumology and Thoracic Surgery (SEPAR) (Unknown); Asociación Española de Afectados de Cáncer de Pulmón (AEACaP) (Unknown); Medtronic General Research Grant (Unknown); Spanish Society of Thoracic Surgery (SECT) (Unknown)
Responsible Party: Sponsor-Investigator, Carlos Alfredo Fraile Olivero, MD, PhD., Principal Investigator, Hospital San Carlos, Madrid
Organization: Hospital San Carlos, Madrid (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 22/310-EC_X
Record Dates: First submitted 2024-11-25; First posted 2024-12-13 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Surgical Procedure, Unspecified; Non Small Cell Lung Cancer; Surgery Scheduled; Thoracic Surgery; Postoperative Complications; Perioperative Care
Keywords: Respiratory physiotherapy; Smartphone App; Post-operative complications; Peri-operative physical training
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Postoperative Complications

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- In-person respiratory physiotherapy (Active Comparator): The patient must attend the respiratory physiotherapy sessions given by physiotherapists at the place and time established in each centre, before and after surgery.
  Interventions: Procedure: On-site respiratory physiotherapy
- Face-to-face respiratory physiotherapy plus use of the Fissios App (Experimental): The same protocol will be followed as for the control group and, in addition, the steps for downloading the application and the start-up will be explained verbally and in writing. The researcher will encourage the patient to use the Fissios App©, read all the perioperative medical recommendations and perform the respiratory physiotherapy exercises freely without restrictions in terms of time, time of use or location.
  Interventions: Procedure: On-site respiratory physiotherapy; Device: Fissios App

INTERVENTIONS:
Procedure: On-site respiratory physiotherapy — The patient attends face-to-face physiotherapy sessions prescribed by the doctor.
Device: Fissios App — The patient uses the Fissios App to perform respiratory physiotherapy exercises.
  Arms: Face-to-face respiratory physiotherapy plus use of the Fissios App

SUMMARY:
Respiratory physiotherapy as part of a pre-operative physical training program may reduce the risk of developing post-operative complications, improving post-operative results and optimizing physical conditions in patients with a diagnosis of non-small cell lung cancer (NSCLC) undergoing lung resection surgery. During the post-operative period, performing physical exercise has also been proved to increase the capacity for exercise, improve health-related quality of life and reduce the feeling of breathlessness. Fissios App is a tool created by thoracic surgeons, physiotherapists and a specialist doctor in physical medicine and rehabilitation, which has been satisfactorily implemented in thoracic surgery patients; this contains a program of standardized respiratory physiotherapy exercises with a defined time and number of repetitions.

The aim is to compare the effectiveness of use of the Fissios App tool as a complement to a peri-operative respiratory physiotherapy program compared to just attendance at a face-to-face peri-operative respiratory physiotherapy program, to reduce the incidence of post-operative complications.

It is expected to include 560 patients in the study. Subsequent to evaluation by the investigator and the acceptance of participant to take part in the study, the performing of peri-operative respiratory physiotherapy is prescribed. The participants will be randomly assigned to a study group that uses the tool as a complement to the respiratory physiotherapy program or a control group that should only attend face-to-face respiratory physiotherapy sessions. All the participants should attend face-to-face respiratory physiotherapy classes taught by physiotherapists at the place and time set out in each centre before and after surgery for at least 45 minutes and at least five sessions. Moreover, study group participants may use the Fissios App tool. Investigators should fill in the pre-operative, surgery and post-operative data for each patient on the Fissios Research platform.

DETAILED DESCRIPTION:
The FPoC Trial is designed as a multicentre, prospective, randomised, prospective, parallel, two-group, controlled, open-label, superiority study of only face-to-face respiratory physiotherapy or the use of Fissios App© as an adjunct to respiratory physiotherapy in patients scheduled for lung resection surgery.

The participants who take part in the study will be randomly assigned to the study or control group before the surgical procedure. All of them will follow an in-person respiratory physiotherapy programme, and the study group will complement this programme with the use of the Fissios App tool.

Perioperative care will be carried out in accordance with national and international guidelines. Postoperative complications will be recorded following the established definitions of the European Society of Thoracic Surgeons (ESTS) database and in the study protocol.

Finally, all the participants will be followed up for 90 days after the date of surgery to finalise the present study. The participants will continue the revisions following the protocols of each centre.

An estimated total of 560 particpants (280 per group) will be recruited for this study.

ELIGIBILITY:
Inclusion Criteria:

1. Patients over 18 years of age.
2. Indication for lung resection surgery due to diagnostic suspicion or histopathological diagnosis of non-small cell lung carcinoma.
3. Anatomical lung resection surgery: anatomical segmental resection, lobectomies or pneumonectomies, using a conventional or minimally invasive approach (VATS, RATS).
4. The patient has a smart mobile device compatible with the Fissios App©, has the ability or has the support to use it.
5. Willingness and commitment to participate in the study.
6. Ability to complete the informed consent to participate in the study.

Exclusion Criteria:

1. Medical contraindication to perform respiratory physiotherapy exercises.
2. Not possessing a smart mobile device compatible with Fissios App©.
3. Inability of the patient to perform the exercises, either due to a physical or psychological impediment.
4. Inability to complete the informed consent form for participation in the study.
5. Refusal to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 560 (Estimated)
Dates: Start 2025-03-20 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Postoperative complications | Through postoperative evolution, an average of 2 weeks.
  Development of at least one adverse clinical event categorised as a postoperative complication during hospital admission. Immediately after the surgery until discharge.

SECONDARY OUTCOMES:
Duration of pleural drainage | Through postoperative evolution, an average of 2 weeks.
  Time that the patient has pleural drainage from the end of surgery until medical discharge.
Mortality | During hospitalization period, an average of 2 weeks.
  Patient status at the moment of discharge.
Hospital readmission | Within 30 days of discharge from hospital
  Any clinical situation requiring hospital admission
Mortality | During the first 30 days after surgery
Mortality | During the first 90 days after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Carlos A Fraile Olivero, MD, PhD, Principal Investigator — Hospital San Carlos, Madrid
Locations (1):
- Hospital Clínico San Carlos, Madrid, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rami-Porta R, Wittekind C, Goldstraw P; International Association for the Study of Lung Cancer (IASLC) Staging Committee. Complete resection in lung cancer surgery: proposed definition. Lung Cancer. 2005 Jul;49(1):25-33. doi: 10.1016/j.lungcan.2005.01.001. PMID 15949587
- [Background] Fernandez FG, Falcoz PE, Kozower BD, Salati M, Wright CD, Brunelli A. The Society of Thoracic Surgeons and the European Society of Thoracic Surgeons general thoracic surgery databases: joint standardization of variable definitions and terminology. Ann Thorac Surg. 2015 Jan;99(1):368-76. doi: 10.1016/j.athoracsur.2014.05.104. PMID 25555970
- [Background] Garutti I, Cabanero A, Vicente R, Sanchez D, Granell M, Fraile CA, Real Navacerrada M, Novoa N, Sanchez-Pedrosa G, Congregado M, Gomez A, Minana E, Pineiro P, Cruz P, de la Gala F, Quero F, Huerta LJ, Rodriguez M, Jimenez E, Puente-Maestu L, Aragon S, Osorio-Salazar E, Sitges M, Lopez Maldonado MD, Rios FT, Morales JE, Callejas R, Gonzalez-Bardancas S, Botella S, Cortes M, Yepes MJ, Iranzo R, Sayas J. Recommendations of the Society of Thoracic Surgery and the Section of Cardiothoracic and Vascular Surgery of the Spanish Society of Anesthesia, Resuscitation and Pain Therapy, for patients undergoing lung surgery included in an intensified recovery program. Rev Esp Anestesiol Reanim (Engl Ed). 2022 Apr;69(4):208-241. doi: 10.1016/j.redare.2021.02.011. Epub 2022 May 15. PMID 35585017
- [Background] Batchelor TJP, Rasburn NJ, Abdelnour-Berchtold E, Brunelli A, Cerfolio RJ, Gonzalez M, Ljungqvist O, Petersen RH, Popescu WM, Slinger PD, Naidu B. Guidelines for enhanced recovery after lung surgery: recommendations of the Enhanced Recovery After Surgery (ERAS(R)) Society and the European Society of Thoracic Surgeons (ESTS). Eur J Cardiothorac Surg. 2019 Jan 1;55(1):91-115. doi: 10.1093/ejcts/ezy301. PMID 30304509
- [Background] Fraile Olivero CA, Jarabo Sarceda JR, Fernandez Martin E, Santos Capa P, Arribas Manzanal PD, Gomez Martinez AM, Calatayud Gastardi J, Hernando Trancho F. Implementation of a perioperative care App in elective thoracic surgery. Cir Esp (Engl Ed). 2023 Apr;101(4):265-273. doi: 10.1016/j.cireng.2022.09.022. Epub 2022 Sep 12. PMID 36108953
- [Background] Rosero ID, Ramirez-Velez R, Lucia A, Martinez-Velilla N, Santos-Lozano A, Valenzuela PL, Morilla I, Izquierdo M. Systematic Review and Meta-Analysis of Randomized, Controlled Trials on Preoperative Physical Exercise Interventions in Patients with Non-Small-Cell Lung Cancer. Cancers (Basel). 2019 Jul 5;11(7):944. doi: 10.3390/cancers11070944. PMID 31284372
- [Background] Mainini C, Rebelo PF, Bardelli R, Kopliku B, Tenconi S, Costi S, Tedeschi C, Fugazzaro S. Perioperative physical exercise interventions for patients undergoing lung cancer surgery: What is the evidence? SAGE Open Med. 2016 Oct 19;4:2050312116673855. doi: 10.1177/2050312116673855. eCollection 2016. PMID 27803808
- [Background] Mans CM, Reeve JC, Elkins MR. Postoperative outcomes following preoperative inspiratory muscle training in patients undergoing cardiothoracic or upper abdominal surgery: a systematic review and meta analysis. Clin Rehabil. 2015 May;29(5):426-38. doi: 10.1177/0269215514545350. Epub 2014 Aug 26. PMID 25160007
- [Background] Kendall F, Oliveira J, Peleteiro B, Pinho P, Bastos PT. Inspiratory muscle training is effective to reduce postoperative pulmonary complications and length of hospital stay: a systematic review and meta-analysis. Disabil Rehabil. 2018 Apr;40(8):864-882. doi: 10.1080/09638288.2016.1277396. Epub 2017 Jan 17. PMID 28093920
- [Background] Cavalheri V, Burtin C, Formico VR, Nonoyama ML, Jenkins S, Spruit MA, Hill K. Exercise training undertaken by people within 12 months of lung resection for non-small cell lung cancer. Cochrane Database Syst Rev. 2019 Jun 17;6(6):CD009955. doi: 10.1002/14651858.CD009955.pub3. PMID 31204439
- [Background] Sebio Garcia R, Yanez Brage MI, Gimenez Moolhuyzen E, Granger CL, Denehy L. Functional and postoperative outcomes after preoperative exercise training in patients with lung cancer: a systematic review and meta-analysis. Interact Cardiovasc Thorac Surg. 2016 Sep;23(3):486-97. doi: 10.1093/icvts/ivw152. Epub 2016 May 25. PMID 27226400
- [Background] Cavalheri V, Granger C. Preoperative exercise training for patients with non-small cell lung cancer. Cochrane Database Syst Rev. 2017 Jun 7;6(6):CD012020. doi: 10.1002/14651858.CD012020.pub2. PMID 28589547